CLINICAL TRIAL: NCT01455545
Title: Impact of Adherence to Treatment in Asthma Control Using ASK-20 Questionnaire and Prescription Account.
Brief Title: Impact of Adherence to Treatment in Asthma Control
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, CARLOS ALMONACID SANCHEZ, PhD, MD, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: HUGU ASMA 001
Record Dates: First submitted 2011-10-10; First posted 2011-10-20 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Asthma; Degree of Control; Exhaled Nitric Oxide; Asthma Control Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This survey aims to analyze how adherence to treatment, using Ask-20 questionnaire and prescription count, influences level of asthma control in a sample of patients with severe and moderate-mild asthma.

DETAILED DESCRIPTION:
Duration of illness, poor adherence to treatment, gender, smoking habit, obesity, concomitant diseases (rhinitis, sinusitis or gastroesophageal reflux) and concomitant psychiatric disorders may be responsible for an increase and perpetuation of the inflammatory response as well as a decreased response to treatment and may be easily identified clinically.

PRIMARY OBJECTIVES: a) analyze how adherence to treatment, using ASK-20 questionnaire and prescription count, influences level of asthma control in a sample of patients with severe and moderate-mild asthma.

SECONDARY OBJECTIVES: a) analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) score and the fraction exhaled of nitric oxide (FeNO); b) analyze the relation between the level of asthma control according to the ACT score and the gender. c) analyze the relation between the level of asthma control according to the ACT score and smoking habit. d) analyze the correlation between the level of asthma control according to the ACT score and obesity. e) analyze the relation between the level of asthma control according to the ACT score and concomitant diseases (rhinitis, sinusitis or gastroesophageal reflux). f) analyze the relation between the level of asthma control according to the ACT score and concomitant psychiatric disorders. g) analyze the relation between the level of asthma control according to the ACT score and disease severity under the terms proposed by Global Initiative for Asthma (GINA).

METHOD: This is a observational cross-sectional study that includes a sample made up of 50 patients with good asthma control and 50 patients with poor asthma control according to the Asthma Control Test(ACT).

DEVELOPMENT OF THE STUDY After signing the informed consent, data will be collected including gender, smoking habit, alcohol consumption, environmental and employment factors, weight, height, body mass index (BMI), history of atopy, disease severity, rhinosinusitis, gastroesophageal reflux and concomitant psychiatric disorders and a standard physical examination. Measurement of asthma control with Asthma Control Test (ACT)will be performed. Then fraction exhaled of nitric oxide (FeNO)measurement and pulmonary function testing (forced spirometry and bronchodilator test) will be performed .

DEVICES AND MEASUREMENTS: Clinical variables will be collected in a case report form (CRF) specially developed for the study. Functional study: The spirometry will be performed according to the recommendations of European Respiratory Society using the Jaeger Master Lab system.

Bronchodilator test will be performed with albuterol and ipratropium bromide inhalation solution. FeNO levels will be measured of using the Filt's Vario analyzer which allows for bronchial or nasal tests, with a flow and volume meter Lilly-type pneumotachograph . Adherence to treatment will be assessed with the ASK-20 questionnaire and reviewing the number of prescriptions for asthma during the last 6 months.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of asthma according to the Global Initiative for Asthma (GINA)guideline criteria .

Exclusion Criteria:

* Patients with a history of chronic obstructive pulmonary disease (COPD), residual pulmonary lesions or bronchiectasis seen on simple chest x-ray.
* Presence of another associated acute or chronic inflammatory disease.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ASTHMA will be categorized into two subgroups: a) 50 patients with good asthma control according to the Asthma Control Test (ACT) score; b) 50 patients with bad control asthma according to the ACT score.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Almonacid Sanchez, Phd, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (1):
- Hospital Universitario de Guadalajara, Guadalajara, Castille-La Mancha, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: Jan 2011 to Jan 2012. Location: medical clinic. Sampling method: Non-Probability Sample. Ages Eligible for Study: 16 yars to 80 years. Genders Eligible for Study: both.
Groups:
- Bad Control: Patient group with bad control defined as participants with an Asthma Control Test (ACT) = or < 19 points.
- Good Control: Patient group with good control defined as participants with an Asthma Control Test (ACT)> 19 points.
Period: Overall Study
Arm/Group | Bad Control | Good Control
Started | 55 | 45
Completed | 55 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asthmatic Patients: Patient group with bad control defined as participants with an Asthma Control Test (ACT) score = or < 19. Patient group with good control defined as participants with an Asthma Control Test (ACT)score > 19.
  In both groups there were patients with mild, moderate and severe asthma according the Global Initiative for Asthma (GINA).
Arm/Group | Asthmatic Patients
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 87
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 45.25 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 34
Region of Enrollment [Number; unit: participants]
  Spain | 100

OUTCOME MEASURES:

1. Primary Outcome: Analyze How Adherence to Treatment Using ASK-20 Questionnaire Influences Level of Asthma Control.
Description: The ASK-20 (Adherence Starts with Knowledge)is a brief, self-reported instrument developed to identify patient-specific barriers to medication adherence and to improve provider/patient communication about adherence.
  Programs incorporating a clinical assessment tool such as the ASK-20 for identifying a broad range of risk factors for nonadherence and for developing patient-specific intervention may reduce adherence barriers and improve disease control and ability to perform daily activities in patients with asthma.
  To gauge the overall risk of nonadherence, the total ASK-20 score was calculated,as the sum of the individual item score, ranging from 1 to 5 and therefore total ranges score from 20 (less barriers to adherence) to 100 (more barriers).
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Bad Control: Patients with asthma and bad control evaluated by Asthma Control Test. Bad control if ACT score < or = 19 .
- Good Control: Patients with asthma and good control evaluated by Asthma Control Test (ACT). Good control if ACT score > 19.
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
units on a scale | 34 [22 to 41] | 32 (15) [22.5 to 43]
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences in ASK-20 results between both groups H1= there are differences between both groups. Comparison of two means. Unilateral test. (1-alpha)=95%. Statistic power: 90%. Precision: 10. S square: 256. Sample size: 44. Sample size adjusted to losses: 46 patients; Test type: Superiority or Other; p = 0.967, Regression, Logistic; Odds Ratio (OR) = 0.999, 95% CI 2-sided [0.962 to 1.037]

2. Secondary Outcome: Fraction Exhaled of Nitric Oxide (FeNO) According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) scores and the fraction exhaled of nitric oxide (FeNO). Units FENO: ppb (parts per billion).
  Asthma control was measured by Asthma Control Test(ACT). Bad control if ACT score < or = 19 . Good control if ACT score > 19.
Time Frame: 4 weeks
Population: The same as primary outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale (parts per billion)
Groups:
- Bad Control: Patients with asthma and bad control evaluated by Asthma Control Test (ACT). Bad control if ACT score < or = 19 .
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
units on a scale (parts per billion) | 27 [17 to 45] | 28 [18.5 to 40]
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Test type: Superiority or Other; p = 0.861, Regression, Logistic; Odds Ratio (OR) = 1.001, 95% CI 2-sided [0.985 to 1.018]

3. Secondary Outcome: Gender According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) scores and the gender.
  Asthma control was measured by Asthma Control Test(ACT). Good control if ACT score > 19. Bad control if ACT score < or = 19.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Good Control: Patients with asthma and good control evaluated by Asthma Control Test. Good control if ACT score > 19.
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  male | 16 | 18
  female | 39 | 27
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences in gender results between both groups H1= there are differences between both groups. Cross tab Chi square; Test type: Superiority or Other; p = 0.252, Chi-squared; Odds Ratio (OR) = 1.625, 95% CI 2-sided [0.706 to 3.739]

4. Secondary Outcome: Smoking Habit According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) score and smoking habit.
  Good control if ACT score > 19. Bad control if ACT score < or = 19. Patients were divided into three types: active smokers, former smokers and people who had never smoked.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Bad Control: Patients with asthma and bad control evaluated by Asthma Control Test. Bad control if ACT score < or = 19.
- Good Control: Patients with asthma and good control evaluated by Asthma Control Test. Good control if ACT score > 19 .
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  current smoker | 7 | 5
  non smoker | 25 | 28
  former smoker | 23 | 12
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Chi - square; Test type: Superiority or Other; p = 0.217, Chi-squared

5. Secondary Outcome: Obesity According to Level of Asthma Control.
Description: Analyze the correlation between the level of asthma control according to the Asthma Control Test (ACT) score and obesity, measured by body mass index(BMI). If BMI (18-25) = normal. If BMI (25 - 29) = overweight. If BMI > 30 obesity.
  Asthma control was measured by Asthma Control test (ACT). Good control if ACT score > 19. Bad control if ACT score < or = 19 .
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  Normal | 28 | 25
  overweight - obesity | 27 | 20
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Cross tabs Chi square; Test type: Superiority or Other; p = 0.643, Chi-squared; Odds Ratio (OR) = 0.830, 95% CI 2-sided [0.376 to 1.829]

6. Secondary Outcome: Rhinitis According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) score and rhinitis.
  Asthma control was measured by Asthma Control Test (ACT). Good control if ACT score > 19. Bad control if ACT score < or = 19.
  Rhinitis was diagnosed by symptoms, according to Allergic Rhinitis and its Impact on Asthma(ARIA)guideline.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Bad Control Asthmatic Patients: Patients with asthma and bad control evaluated by Asthma Control Test (ACT). Bad control if ACT score < or = 19.
Arm/Group | Bad Control Asthmatic Patients | Good Control
Number analyzed (Participants) | 55 | 45
participants
  yes | 18 | 21
  no | 37 | 24
Statistical Analysis 1: Comparison: Bad Control Asthmatic Patients vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Cross tabs Chi squared test; Test type: Superiority or Other; p = 0.155, Chi-squared; Odds Ratio (OR) = 0.556, 95% CI 2-sided [0.247 to 1.253]

7. Secondary Outcome: Sinusitis According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) Score and Sinusitis.
  Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19. Good control if ACT score > 19.
  Diagnosis of sinusitis was established according to The European Position Paper on Rhinosinusitis and Nasal Polyps (EP3OS) group.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Bad Control Asthmatic Patients: Patients with asthma and bad control evaluated by Asthma Control Test. Bad control if ACT score < or = 19.
Arm/Group | Bad Control Asthmatic Patients | Good Control
Number analyzed (Participants) | 55 | 45
participants
  yes | 1 | 4
  no | 54 | 41
Statistical Analysis 1: Comparison: Bad Control Asthmatic Patients vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Cross tabs Chi squared test; Test type: Superiority or Other; p = 0.107, Chi-squared; Odds Ratio (OR) = 0.190, 95% CI 2-sided [0.020 to 1.763]

8. Secondary Outcome: Gastroesophageal Reflux According to Level of Asthma Control.
Description: Analyze the relation Between the Level of Asthma Control According to the ACT Score and gastroesophageal reflux.
  Gastroesophageal reflux was diagnosed by symptoms or previous diagnosis in their medical records with or without treatment for reflux.
  Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19. Good control if ACT score > 19.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Bad Control: Patients with asthma and bad control. Bad control if ACT score < or = 19.
- Good Control: Patients with asthma and goog control. Good control if ACT score > 19.
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 44
participants
  yes | 2 | 0
  no | 53 | 45
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Cross tabs Chi squared test; Test type: Superiority or Other; p = 0.196, Chi-squared; Odds Ratio (OR) = 1.849, 95% CI 2-sided [1.541 to 2.219]

9. Secondary Outcome: Concomitant Psychiatric Disorders According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the Asthma Control Test (ACT) score and concomitant psychiatric disorders.
  Depression and anxiety were the concomitant psychiatric disorders. Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19. Good control if ACT score > 19.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  yes | 7 | 2
  no | 48 | 43
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Cross tabs Chi squared test; Test type: Superiority or Other; p = 0.150, Chi-squared; Odds Ratio (OR) = 3.135, 95% CI 2-sided [0.618 to 15.91]

10. Primary Outcome: Analyze How Adherence to Treatment Using Prescription Account Influences Level of Asthma Control.
Description: Analyze how adherence to treatment using prescription count influences level of asthma control in a sample of patients with severe and moderate-mild asthma. The second primary endpoint analyzes how adherence, using prescription counts, influences the level of asthma control. Good adherence to treatment was defined as a count of prescriptions issued by their family physician greater than 80% of the required treatment during the last 6 months.
  Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19 . Good control if ACT score > 19.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Good Control: Patients with asthma and good control evaluated by Asthma Control Test (ACT). Good control if ACT score > 19 .
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  adherence to inhalers >= 80% | 33 | 26
  adherence to inhalers < 80% | 22 | 19
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups. Comparison of two proportions. Unilateral test. (1-alpha)=95%. Proportion: 90%. Precision: 10%. Sample size: 35. Sample size adjusted to losses: 41 patients; Test type: Superiority or Other; p = 0.822, Chi-squared; Odds Ratio (OR) = 1.096, 95% CI 2-sided [0.492 to 2.441]

11. Secondary Outcome: Pulmonary Function Test (Spirometry) According to Level of Asthma Control.
Description: Analyze the relation between the level of asthma control according to the ACT scores and pulmonary function test (spirometry).
  Functional study. The Master Lab system (Jaeger, Wurzburg, Germany) was used to obtain spirometry parameters Respiratory function tests were performed according to the recommendations of the European Respiratory Society. The predicted values used for pulmonary function variables were obtained from the European Community for Coal and Steel. This will be performed according to the recommendations of European Respiratory Society using the Jaeger Master Lab system.
  Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19. Good control if ACT score > 19.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of the theoretical
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
percentage of the theoretical | 84.23 (16.49) | 94.93 (18.04)
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Bad Control vs Good Control; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 1.038, 95% CI 2-sided [1.012 to 1.065]

12. Secondary Outcome: Asthma Severity According to Level of Asthma Control.
Description: Analyze the relation Between the Level of Asthma Control According to the Asthma Control Test (ACT) Score and asthma severity according the Global Initiative for Asthma (GINA).
  Asthma control was measured by Asthma Control Test (ACT). Bad control if ACT score < or = 19. Good control if ACT score > 19.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Bad Control | Good Control
Number analyzed (Participants) | 55 | 45
participants
  mild-moderate asthma | 24 | 31
  severe asthma | 31 | 14
Statistical Analysis 1: Comparison: Bad Control vs Good Control; Ho = no differences between both groups H1= there are differences between both groups; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 0.350, 95% CI 2-sided [0.153 to 0.799]

ADVERSE EVENTS:
Time Frame: This is a cross-sectional study in which all data are collected in a single visit. There is no treatment previously modified or new drugs were tested. No intervention was performed so it can not be collected any adverse effects.
Groups:
- Bad Control Asthmatic Patients: Patients with asthma and bad control evaluated by Asthma Control Test. Good control less than 20 score.
- Good Control: Patients with asthma and good control evaluated by Asthma Control Test. Good control more than 19 score.
Arm/Group | Bad Control Asthmatic Patients | Good Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This is an observational (cross-sectional )study, with the limitations and biases associated. Patients have not been randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes